CLINICAL TRIAL: NCT02928874
Title: Eating Phenotypes for Childhood Obesity in the Context of Familial Obesity Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 820661
Record Dates: First submitted 2016-10-04; First posted 2016-10-10 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Caloric compensation (Experimental): Twenty-five minutes before breakfast, participants will be asked to consume in full one of two oatmeal preloads that will vary in ED. The order of preload conditions will be randomized across groups of children participating in the visits.
  Interventions: Behavioral: % COMPX (low ED vs. high ED preload)
- Eating in the absence of hunger (EAH) (Experimental): During both study visits, children's EAH will be assessed after lunch and again after dinner. The order of presenting the low and high ED snacks will be counterbalanced across meals.
  Interventions: Behavioral: EAH (low ED vs. high ED snacks)

INTERVENTIONS:
Behavioral: % COMPX (low ED vs. high ED preload)
  Arms: Caloric compensation
Behavioral: EAH (low ED vs. high ED snacks)
  Arms: Eating in the absence of hunger (EAH)

SUMMARY:
Using an integrated approach, this study examines multiple eating traits concurrently under states of hunger and satiety. It examines the impact of short-term appetite and intake regulation on longer-term energy intake control and weight development in a cohort of ethnically diverse normal-weight and obese boys and girls with different familial predispositions to obesity.

ELIGIBILITY:
Inclusion Criteria:

* 7-9 years of age
* Normal-weight or overweight/obese who are at low risk or high risk for obesity based on maternal BMI
* Like most foods served during the study
* Be regular breakfast eaters

Exclusion Criteria:

* Have serious medical conditions known to affect food intake or body weight
* Have any developmental, medical, or psychiatric conditions that might impact study compliance
* Have a learning disability or poor reading ability/comprehension
* Have visual or auditory impairment
* Are taking medications associated with developmental, medical, or psychiatric disorders or medications known to affect appetite, food intake or body weight
* Are underweight
* Have food allergies related to the foods served in the study or are lactose intolerant
* Do not regularly eat breakfast
* Do not like or cannot eat foods served during experimental meal or are unable to finish compulsory preload
* Mothers who are pregnant

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Percent caloric compensation index (%COMPX) | Baseline
Appetite ratings assessed via Visual Analog Scales | Baseline
  Appetite ratings include self-reported perceived hunger, desire to eat, prospective consumption, and fullness.
Total energy intake per day (number of calories consumed over 24-hours) | Baseline
  Number of calories consumed over 24-hours assessed via measured food intake in the laboratory and via parent-reported food intake at home.
BMI z-score | Change from baseline BMI z-score at 1-year follow-up
Waist circumference (cm) | Change from baseline waist circumference at 1-year follow-up
Percentage body fat | Change from baseline percentage body fat at 1-year follow-up

SECONDARY OUTCOMES:
Eating in the absence of hunger (kcal) | Baseline (number of calories consumed from snacks)
Home food environment | Baseline home food environment assessed using the Home Food Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Kral, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kral TVE, Moore RH, Chittams J, O'Malley L, Jones E, Quinn RJ, Fisher JO. Caloric compensation and appetite control in children of different weight status and predisposition to obesity. Appetite. 2020 Aug 1;151:104701. doi: 10.1016/j.appet.2020.104701. Epub 2020 Apr 11. PMID 32289325